CLINICAL TRIAL: NCT03417674
Title: SHAPE AND MOTION - Medical Accompanied Slimming
Acronym: SAMMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: FORM UND BEWEGUNG
Record Dates: First submitted 2018-01-09; First posted 2018-01-31 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Lifestyle intervention with meal replacement by formula diet, exercise stimulation, and telemedicine coaching.
  Interventions: Combination Product: Lifestyle intervention
- Control group (No Intervention): Routine care.

INTERVENTIONS:
Combination Product: Lifestyle intervention — Meal replacement by formula diet, exercise stimulation, and telemedicine coaching.
  Arms: Intervention group

SUMMARY:
Background: Overweight and obesity affect health, quality of life and ability to work. Therefore, the scientifically evaluated program "SHAPE AND MOTION - medically ◦ accompanied ◦ slimming" was developed to support overweight and obese people in weight loss.

Method: In a randomized controlled clinical trial, the effect of a lifestyle intervention with meal replacement by formula diet, exercise stimulation, and telemedicine coaching is examined compared to a control group with routine care. The learning contents are taught in 7 group trainings, a practical unit with shopping and cooking training, as well as in 4 individual telephone conversations. The state of health is examined at the beginning, after 12 and 26 weeks.

Objective: The aim is to develop a training and counseling program for overweight or obese individuals with diabetes risk or type 2 diabetes, which can be used both for primary and for tertiary prevention of overweight-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 25 kg/m2

Exclusion Criteria:

* acute diseases such as respiratory or gastrointestinal infections
* severe diseases such as tumors, chronic obstructive pulmonary disease (COPD), asthma, dementia, chronic bowel disease, psychosis, liver cirrhosis, (macro) nephropathy, renal insufficiency with glomerular filtration rate (GFR) <30
* ongoing chemotherapy, chron. Cortisone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Weight loss in kg | 26 weeks
  Estimated treatment difference

SECONDARY OUTCOMES:
body mass index in kg/m2 | 26 weeks
  Estimated treatment difference
waist circumference in cm | 26 weeks
  Estimated treatment difference
hip circumference in cm | 26 weeks
  Estimated treatment difference
fat mass in kg | 26 weeks
  Estimated treatment difference
lean body mass in kg | 26 weeks
  Estimated treatment difference
muscle mass in kg | 26 weeks
  Estimated treatment difference
energy expenditure in kcal | 26 weeks
  Estimated treatment difference
blood pressure in mmHg | 26 weeks
  Estimated treatment difference
quality of life (sf-12 questionnaire) in units on a scale | 26 weeks
  Estimated treatment difference
depression (German version of the Center for Epidemiological Studies-Depression [CES-D] Scale) in units on a scale | 26 weeks
  Estimated treatment difference
physical activity in min/day | 26 weeks
  Estimated treatment difference
physical activity in steps/day | 26 weeks
  Estimated treatment difference
eating behaviour (German version of the Three-factor Eating Questionnaire [TFEQ]) in units on a scale | 26 weeks
  Estimated treatment difference
total cholesterol in mg/dl | 26 weeks
  Estimated treatment difference
HDL cholesterol in mg/dl | 26 weeks
  Estimated treatment difference
LDL cholesterol in mg/dl | 26 weeks
  Estimated treatment difference
triglycerides in mg/dl | 26 weeks
  Estimated treatment difference
fasting blood glucose in mg/dl | 26 weeks
  Estimated treatment difference
insulin in µU/ml | 26 weeks
  Estimated treatment difference
HbA1c in % | 26 weeks
  Estimated treatment difference
uric acid in mg/dl | 26 weeks
  Estimated treatment difference
creatinin in mg/dl | 26 weeks
  Estimated treatment difference
medication in mg/day | 26 weeks
  Estimated treatment difference

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West-German Centre of Diabetes and Health
Locations (1):
- West-German Centre of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No